CLINICAL TRIAL: NCT01102426
Title: Randomized, Multicenter, Open-label, Phase III Study of Plitidepsin in Combination With Dexamethasone vs. Dexamethasone Alone in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Aplidin - Dexamethasone in Relapsed/Refractory Myeloma
Acronym: ADMYRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APL-C-001-09
Record Dates: First submitted 2010-03-31; First posted 2010-04-13 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Relapsed/Refractory Multiple Myeloma
Keywords: Multiple Myeloma; Aplidin; plitidepsin; dexamethasone
MeSH Terms: conditions — Multiple Myeloma | interventions — plitidepsin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Plitidepsin+Dexamethasone (Experimental): plitidepsin + dexamethasone combination
  Interventions: Drug: Plitidepsin; Drug: Dexamethasone
- Dexamethasone (Active Comparator): dexamethasone single agent
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Plitidepsin — plitidepsin: powder and solvent for concentrate for solution for infusion. 2 mg vial + 4 ml ampoule. 5 mg/m2 intravenously (i.v.) over three hours on Day 1 and 15 every 4 weeks. dexamethasone: 4 mg tablet. 40 mg orally on Day 1, 8, 15 and 22 every four weeks at least one hour before plitidepsin infusion.
  Other Names: APLIDIN (plitidepsin)
  Arms: Plitidepsin+Dexamethasone
Drug: Dexamethasone — 4 mg tablet. 40 mg orally on Day 1, 8, 15 and 22 every four weeks.
  Other Names: DXN

SUMMARY:
Study of Plitidepsin in combination with dexamethasone versus dexamethasone alone in patients with relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
Phase III Study in Patients with Relapsed/Refractory Multiple Myeloma to compare the efficacy of plitidepsin in combination with dexamethasone vs. dexamethasone alone measured by progression-free survival (PFS) and to evaluate tumor response, duration of response (DR), overall survival (OS) and to rule out any effect of plitidepsin on the duration of the QT/QTc interval (time corresponding to the beginning of depolarization to re-polarization of the ventricles).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤ 2
* Life expectancy ≥ 3 months.
* Patients previously diagnosed with multiple myeloma
* Patients must have relapsed or relapsed and refractory multiple myeloma (MM) after at least three but not more than six prior therapeutic regimens for MM, including induction therapy and stem cell transplant in candidate patients, which will be considered as only one regimen.
* Patients must have received previous bortezomib-containing and lenalidomide-containing regimens (or thalidomide where lenalidomide is not available)
* Women must have a negative serum pregnancy test
* Voluntarily signed and dated written informed consent

Exclusion Criteria:

* Concomitant diseases/conditions
* Women who are pregnant or breast feeding.
* Concomitant medications that include corticosteroids, chemotherapy, or other therapy that is or may be active against MM
* Known hypersensitivity to any involved study drug or any of its formulation components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2010-06; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Óscar F. Ballester, M.D., Principal Investigator — Edwards Comprehensive Cancer Center, Marshall University (Huntington); Rubén Niesvizky, M.D., Principal Investigator — NY Presbyterian Hosp. - Cornell University - NY
Locations (82):
- United States (5):
  - 1107, Tuscaloosa, Alabama
  - 1103, Los Angeles, California
  - 1105, Jacksonville, Florida
  - 1102, New York, New York
  - 1104, Canton, Ohio
- Australia (7):
  - 108, Adelaide
  - 102, Canberra
  - 101, Geelong
  - 105, Parkville
  - 106, Perth
  - 104, South Brisbane
  - 109, Woodville
- Austria (6):
  - 202, Graz
  - 204, Innsbruck
  - 203, Salzburg
  - 201, Vienna
  - 205, Vienna
  - 208, Vienna
- Belgium (4):
  - 304, Bruges
  - 301, Brussels
  - 303, Brussels
  - 302, Ghent
- Czechia (3):
  - 502, Brno
  - 503, Hradec Králové
  - 501, Prague
- France (4):
  - 601, Lille
  - 602, Nantes
  - 606, Rouen
  - 604, Vandœuvre-lès-Nancy
- Germany (8):
  - 709, Düsseldorf
  - 705, Essen
  - 706, Frankfurt
  - 707, Frankfurt
  - 708, Freiburg im Breisgau
  - 703, Heidelberg
  - 702, München
  - 704, Würzburg
- Greece (3):
  - 1301, Athens
  - 1303, Pátrai
  - 1302, Thessaloniki
- 1401, Dublin, Ireland
- Italy (6):
  - 806, Bari
  - 801, Genova
  - 805, Reggio Emilia
  - 803, Rozzano
  - 804, San Giovanni Rotondo
  - 802, Torino
- Netherlands (2):
  - 901, Rotterdam
  - 902, Rotterdam
- New Zealand (2):
  - 1601, Christchurch
  - 1602, Takapuna
- Poland (2):
  - 1704, Opole
  - 1703, Warsaw
- Portugal (2):
  - 1802, Braga
  - 1801, Porto
- 2001, San Juan, Puerto Rico
- South Korea (9):
  - 1502, Anyang
  - 1501, Daejeon
  - 1507, Hwasun
  - 1506, Incheon
  - 1505, Jeonju
  - 1508, Seongnam
  - 1503, Seoul
  - 1504, Seoul
  - 1509, Seoul
- Spain (10):
  - 1201, Barcelona
  - 1203, Barcelona
  - 1209, Barcelona
  - 1207, Madrid
  - 1210, Madrid
  - 1206, Murcia
  - 1204, Palma de Mallorca
  - 1208, Salamanca
  - 1202, San Sebastián
  - 1205, Valencia
- Taiwan (3):
  - 1901, Taipei
  - 1902, Taipei
  - 1903, Taipei
- United Kingdom (4):
  - 1003, Bournemouth
  - 1004, Bradford
  - 1001, London
  - 1005, Nottingham

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 255 patients were enrolled. 171 Group A (Plitidepsin in combination with DXM) and 84 Group B (DXM alone).
  Enrolled patients between 29Jun10 and 19May15 (Last randomization). The first dose of the first patient was given on 19May15 and the last dose of the last patient was given on 07Aug17.
Groups:
- Plitidepsin+Dexamethasone: plitidepsin + dexamethasone combination
  plitidepsin + dexamethasone: plitidepsin: powder and solvent for concentrate for solution for infusion. 2 mg vial + 4 ml ampoule. 5 mg/m2 intravenously (i.v.) over three hours on Day 1 and 15 every 4 weeks. dexamethasone: 4 mg tablet. 40 mg orally on Day 1, 8, 15 and 22 every four weeks at least one hour before plitidepsin infusion.
Period: Overall Study
Arm/Group | Plitidepsin+Dexamethasone | Dexamethasone
Started | 171 | 84
Completed | 6 | 3
Not Completed | 165 | 81
Not completed — Randomized but not treated | 4 | 1
Not completed — Adverse Events (treatment-related) | 15 | 8
Not completed — Physician Decision | 9 | 6
Not completed — Progressive Disease | 85 | 44
Not completed — Adverse Events (unrelated to | 9 | 1
Not completed — Patient Refusal | 24 | 12
Not completed — Death (due to adverse events | 0 | 1
Not completed — Death (non-related to the study | 19 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Plitidepsin+Dexamethasone | Dexamethasone | Total
Number analyzed (Participants) | 171 | 84 | 255
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 88 | 36 | 124
  >=65 years | 83 | 48 | 131
Age, Continuous [Median (Full Range); unit: years] | 64 [36 to 85] | 65 [42 to 85] | 65 [36 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 49 | 123
  Male | 97 | 35 | 132
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 1 | 7
  Czechia | 23 | 10 | 33
  United Kingdom | 12 | 6 | 18
  Portugal | 2 | 1 | 3
  Spain | 13 | 7 | 20
  Greece | 12 | 7 | 19
  New Zealand | 7 | 1 | 8
  Austria | 21 | 7 | 28
  South Korea | 8 | 4 | 12
  Netherlands | 5 | 4 | 9
ECOG PS [Count of Participants; unit: Participants] — ECOG PS, Eastern Cooperative Oncology Group performance status PS 0 Fully active, able to carry on all pre-disease performance without restriction PS 1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature PS 2 Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours PS 3 Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours PS 4 Completely disabled; cannot carry on any selfcare; totally confined to bed or chair PS 5 Dead
  Participants
    PS 0 | 68 | 31 | 99
    PS 1 | 74 | 42 | 116
    PS 2 | 28 | 11 | 39
    PS 3 | 1 | 0 | 1
MM type at diagnosis [Count of Participants; unit: Participants]
  Non Secretory | 6 | 1 | 7
  Secretory IgA | 35 | 21 | 56
  Secretory IgD | 1 | 1 | 2
  Secretory IgG | 101 | 51 | 152
  Secretory IgM | 1 | 0 | 1
  Secretory Light chain disease | 27 | 10 | 37
Durie-Salmon stage at diagnosis [Count of Participants; unit: Participants] — Stage I: small number of myeloma cells. All are present:Hemoglobin>100 g/L;Blood calcium<2.8 mmol/L;No areas of bone damage or a solitary plasmacytoma of the bone;IgG<50 g/L;IgA<30 g/L;Urine M-protein<4 g Stage II: Moderate number of myeloma cells. The features are between stage 1 and 3 Stage III: Large number of myeloma cells. One/more are present: Hemoglobin<85 g/L;Blood calcium>2.8 mmol/L;Several areas of bone damage;IgG>70 g/L;IgA>50 g/L;Urine M-protein>12 g Substage A: Kidney function is normal. Creatinine<180 µmol/L. Substage B: Kidney function is abnormal. Creatinine>=180 µmol/L
  Participants
    Stage A | 0 | 1 | 1
    Stage IA | 21 | 9 | 30
    Stage IB | 0 | 2 | 2
    Stage II | 3 | 1 | 4
    Stage IIA | 44 | 20 | 64
    Stage IIB | 1 | 0 | 1
    Stage III | 2 | 1 | 3
    Stage IIIA | 85 | 43 | 128
    Stage IIIB | 14 | 7 | 21
    Not Durie-Salmon stage at diagnosis | 1 | 0 | 1
International Staging System at diagnosis [Count of Participants; unit: Participants] — The International Staging System uses the results of 2 blood tests: albumin and beta-2-microglobulin level.
  Stage I: Beta-2-microglobulin level less than 3.5 mg/L and albumin level more equal than 35 g/L.
  Stage II: Beta-2-microglobulin level less than 3.5 mg/L and Albumin level less than 35 g/L or beta-2-microglobulin level is more than 3.5 mg/L but less than 5.5 mg/L and any albumin level.
  Stage III: Beta-2-microglobulin is 5.5 mg/L or more and any albumin level.
  Participants
    Stage I | 72 | 33 | 105
    Stage II | 41 | 18 | 59
    Stage III | 23 | 15 | 38
    Not stage at diagnosis | 35 | 18 | 53
Cytogenetic risk group at diagnosis [Count of Participants; unit: Participants] — NA: not available; ND: not done; UK: unknown.
  Participants
    Standard risk | 34 | 21 | 55
    High risk | 38 | 16 | 54
    NA/ND/UK | 99 | 47 | 146
Prior radiotherapy [Count of Participants; unit: Participants]
  Yes | 68 | 35 | 103
  No | 103 | 49 | 152
Hb [Median (Full Range); unit: g/dL] | 10.4 [7 to 14.6] | 10.1 [7.4 to 14.6] | 10.3 [7 to 14.6]
Platelets [Median (Full Range); unit: platelets*10^9/L] | 140 [11 to 517] | 154 [24 to 452] | 144 [11 to 517]
CrCL [Median (Full Range); unit: mL/min] — creatinine clearance
  mL/min | 72.9 [21.9 to 252.2] | 69.4 [23 to 137] | 71.9 [21.9 to 252.2]
Time from first diagnosis to randomization [Median (Full Range); unit: months] | 71.8 [0.1 to 277.2] | 70 [19.5 to 178.9] | 71.3 [0.1 to 277.2]
Time from last PD/relapse to first study dose [Median (Full Range); unit: weeks] — PD, Progressive disease .
  weeks | 6.1 [-0.4 to 83.1] | 6.4 [1.0 to 101.7] | 6.2 [-0.4 to 101.7]
Beta-2 microglobulin [Median (Full Range); unit: mg/L] | 4.1 [0.0 to 27.3] | 4.2 [0.2 to 65] | 4.1 [0.0 to 65]
Number of lines of prior systemic therapy [Median (Inter-Quartile Range); unit: lines] | 4 [2 to 6] | 4 [3 to 7] | 4 [2 to 7]

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) as Per Intention-to-treat (ITT)
Description: To compare the efficacy of plitidepsin in combination with dexamethasone vs. dexamethasone alone as measured by progression-free survival (PFS) in patients with relapsed/refractory multiple myeloma (MM).
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Plitidepsin+Dexamethasone | Dexamethasone
Number analyzed (Participants) | 171 | 84
months | 2.6 [1.9 to 3.0] | 1.7 [1.1 to 2.0]
Statistical Analysis 1: Comparison: Plitidepsin+Dexamethasone vs Dexamethasone; Test type: Superiority; p = 0.0054, Log Rank — Cox regression: HR p=0.0062; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.447 to 0.885]

2. Primary Outcome: Percentage of Participants With Progression Free Survival (PFS) as Per Intention-to-treat (ITT) at 6 Months
Description: as for outcome 1
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Plitidepsin+Dexamethasone | Dexamethasone
Number analyzed (Participants) | 171 | 84
percentage of participants | 20.0 [13.1 to 26.9] | 10.0 [2.0 to 18.0]
Statistical Analysis 1: Comparison: Plitidepsin+Dexamethasone vs Dexamethasone; Test type: Superiority; p = 0.0618, Normal approximation

3. Secondary Outcome: Progression-free Survival (Investigator Assessment)
Description: The secondary study analysis was based on Investigator's assessment PFS data in the ITT efficacy population, defined as all patients randomized to either treatment arm. PFS was calculated from randomization to the first evidence of PD or death due to any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions If the patient received further antitumor therapy before PD and within the timeframe expected for first follow-up, PFS was censored on the date of the last disease assessment prior to the administration of this antitumor therapy.
Time Frame: as for outcome 1
Population: All Randomized Patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Plitidepsin+Dexamethasone | Dexamethasone
Number analyzed (Participants) | 171 | 84
months | 2.9 [2.1 to 3.7] | 1.1 [1.0 to 1.9]
Statistical Analysis 1: Comparison: Plitidepsin+Dexamethasone vs Dexamethasone; Test type: Superiority; p < 0.0001, Log Rank — Cox regression HR: p<0.0001; Hazard Ratio (HR) = 0.512, 95% CI 2-sided [0.382 to 0.686]

4. Secondary Outcome: Percentage of Participants With Progression-free Survival (Investigator Assessment) at 6 Months
Description: as for outcome 3
Time Frame: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Plitidepsin+Dexamethasone | Dexamethasone
Number analyzed (Participants) | 171 | 84
percentage of participants | 26.4 [19.1 to 33.7] | 8.1 [1.9 to 14.3]
Statistical Analysis 1: Comparison: Plitidepsin+Dexamethasone vs Dexamethasone; Test type: Superiority; p = 0.0002, Normal approximation

5. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) is defined as the time from the date of randomization to the date of death or last contact
Time Frame: From randomization to the death due to any cause,assessed up to 5 years
Population: All Randomized Patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Plitidepsin+Dexamethasone | Dexamethasone
Number analyzed (Participants) | 171 | 84
months | 11.6 [9.2 to 16.1] | 8.9 [6.0 to 15.4]
Statistical Analysis 1: Comparison: Plitidepsin+Dexamethasone vs Dexamethasone; Pre-specified; Test type: Superiority; p = 0.1261, Log Rank — Cox regression HR: p=0.1273; Hazard Ratio (HR) = 0.797, 95% CI 2-sided [0.596 to 1.067]

6. Secondary Outcome: Percentage of Participants With Overall Survival at 12 Months
Description: Overall Survival (OS) is defined as the time from the date of randomization to the date of death or last contact
Time Frame: From randomization to the death due to any cause,assessed up to 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Plitidepsin+Dexamethasone | Dexamethasone
Number analyzed (Participants) | 171 | 84
percentage of participants | 48.3 [40.4 to 56.2] | 42.1 [31.3 to 52.9]
Statistical Analysis 1: Comparison: Plitidepsin+Dexamethasone vs Dexamethasone; Test type: Superiority; p = 0.3625, Normal approximation

7. Secondary Outcome: Percentage of Participants With Overall Survival at 24 Months
Description: Overall Survival (OS) is defined as the time from the date of randomization to the date of death or last contact
Time Frame: From randomization to the death due to any cause,assessed up to 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Plitidepsin+Dexamethasone | Dexamethasone
Number analyzed (Participants) | 171 | 84
percentage of participants | 30.8 [23.3 to 38.3] | 21.0 [12.0 to 30.1]
Statistical Analysis 1: Comparison: Plitidepsin+Dexamethasone vs Dexamethasone; Test type: Superiority; p = 0.1037, Normal approximation

8. Secondary Outcome: Duration of Response (Independent Review Committee)
Description: DR was calculated from the date of first documentation of response to the date of disease progression or death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From the date of first documentation of response to the date of disease progression or death, assessed up to 5 years
Population: Patients with documentation of response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Plitidepsin+Dexamethasone | Dexamethasone
Number analyzed (Participants) | 39 | 3
months | 3.7 [2.7 to 10.5] | 1.8 [1.8 to 5.5]
Statistical Analysis 1: Comparison: Plitidepsin+Dexamethasone vs Dexamethasone; Test type: Superiority; p = 0.1015, Log Rank — Cox regression HR: 0.1247; Hazard Ratio (HR) = 0.384, 95% CI 2-sided [0.113 to 1.303]

9. Secondary Outcome: Percentage of Participants With Duration of Response (Independent Review Committee) at 6 Months
Description: as for outcome 8
Time Frame: From the date of first documentation of response to the date of disease progression or death, assessed up to 6 months
Population: Patients with documentation of response
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Plitidepsin+Dexamethasone | Dexamethasone
Number analyzed (Participants) | 39 | 3
percentage of participants | 41.2 [24.6 to 57.7] | 0.0 [0.0 to NA] — not reached

10. Secondary Outcome: Duration of Response (Investigator Assessment)
Description: as for outcome 8
Time Frame: From the date of first documentation of response to the date of disease progression or death, assessed up to 5 years
Population: Patients with documentation of response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Plitidepsin+Dexamethasone | Dexamethasone
Number analyzed (Participants) | 51 | 1
months | 5.1 [3.2 to 6.2] | 0.9 [NA to NA] — not reached
Statistical Analysis 1: Comparison: Plitidepsin+Dexamethasone vs Dexamethasone; Pre-specified; Test type: Superiority; p = 0.0001, Log Rank — Cox regression HR: 0.0105; Hazard Ratio (HR) = 0.043, 95% CI 2-sided [0.004 to 0.479]

11. Secondary Outcome: Percentage of Participants With Duration of Response (Investigator Assessment) at 6 Months
Description: as for outcome 8
Time Frame: From the date of first documentation of response to the date of disease progression or death, assessed up to 6 months
Population: Patients with documentation of response
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Plitidepsin+Dexamethasone | Dexamethasone
Number analyzed (Participants) | 51 | 1
percentage of participants | 38.2 [23.7 to 52.8] | 0.0 [0.0 to NA] — not reached

12. Secondary Outcome: Best Overall Response (Independent Review Committee)
Description: Very good partial response (VGPR) serum and urine M-protein detectable but not electrophoresis or >90% reduction in serum M-protein and urine M-protein <100 mg/24h Partial response (PR) ≥50% reduction in serum M-protein and 90% reduction in 24h urine M-protein or to <200 mg/24h. 50% reduction in size of any soft tissue plasmacytomas Minor response (MR) 25%-49% reduction of serum M-protein and 50-89% reduction of 24h urine M-protein. 25-49% reduction in size of soft tissue plasmacytomas. No increase in size or number of bone lesions Stable disease (SD) No sCR, CR, VGPR, PR, MR or PD Progressive disease (PD) 25% increase from the lowest value: serum M-protein, urine M-protein, BM plasma cell. Increase in size, new bone lesions, soft tissue plasmacytomas or serum calcium >11.5 mg/dL; NE, not evaluable
Time Frame: From the date of first documentation of response to the date of disease progression or death, assessed up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Plitidepsin+Dexamethasone | Dexamethasone
Number analyzed (Participants) | 171 | 84
Participants
  VGR | 2 | 0
  PR | 15 | 1
  MR | 22 | 2
  SD | 43 | 21
  PD | 41 | 35
  NE | 48 | 25

13. Secondary Outcome: Overall Response Rate (Independent Review Committee)
Description: Overall response rate including sCR, CR, VGPR, PR and MR. Very good partial response (VGPR) serum and urine M-protein detectable but not electrophoresis or >90% reduction in serum M-protein and urine M-protein <100 mg/24h Partial response (PR) ≥50% reduction in serum M-protein and 90% reduction in 24h urine M-protein or to <200 mg/24h. 50% reduction in size of any soft tissue plasmacytomas Minor response (MR) 25%-49% reduction of serum M-protein and 50-89% reduction of 24h urine M-protein. 25-49% reduction in size of soft tissue plasmacytomas. No increase in size or number of bone lesions
Time Frame: From the date of first documentation of response to the date of disease progression or death, assessed up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Plitidepsin+Dexamethasone | Dexamethasone
Number analyzed (Participants) | 171 | 84
percentage of participants | 22.8 [16.8 to 29.8] | 3.6 [0.7 to 10.1]
Statistical Analysis 1: Comparison: Plitidepsin+Dexamethasone vs Dexamethasone; Test type: Superiority; p < 0.0001, Fisher Exact

14. Secondary Outcome: Overall Response Rate (Independent Review Committee) Excluding MR
Description: Includes sCR, CR, VGPR and PR (excludes MR). Very good partial response (VGPR) serum and urine M-protein detectable but not electrophoresis or >90% reduction in serum M-protein and urine M-protein <100 mg/24h Partial response (PR) ≥50% reduction in serum M-protein and 90% reduction in 24h urine M-protein or to <200 mg/24h. 50% reduction in size of any soft tissue plasmacytomas
Time Frame: From the date of first documentation of response to the date of disease progression or death, assessed up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Plitidepsin+Dexamethasone | Dexamethasone
Number analyzed (Participants) | 171 | 84
percentage of participants | 9.9 [5.9 to 15.4] | 1.2 [0.03 to 6.5]
Statistical Analysis 1: Comparison: Plitidepsin+Dexamethasone vs Dexamethasone; Test type: Superiority; p = 0.0085, Fisher Exact

15. Secondary Outcome: Best Overall Response (Investigator Assessment)
Description: as for outcome 12
Time Frame: From the date of first documentation of response to the date of disease progression or death, assessed up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Plitidepsin+Dexamethasone | Dexamethasone
Number analyzed (Participants) | 171 | 84
Participants
  VGPR | 4 | 0
  PR | 16 | 1
  MR | 31 | 0
  SD | 61 | 31
  PD | 37 | 39
  NE | 22 | 13

16. Secondary Outcome: Overall Response Rate (Investigator Assessment)
Description: Includes sCR, CR, VGPR, PR and MR. Very good partial response (VGPR) serum and urine M-protein detectable but not electrophoresis or >90% reduction in serum M-protein and urine M-protein <100 mg/24h Partial response (PR) ≥50% reduction in serum M-protein and 90% reduction in 24h urine M-protein or to <200 mg/24h. 50% reduction in size of any soft tissue plasmacytomas Minor response (MR) 25%-49% reduction of serum M-protein and 50-89% reduction of 24h urine M-protein. 25-49% reduction in size of soft tissue plasmacytomas. No increase in size or number of bone lesions
Time Frame: From the date of first documentation of response to the date of disease progression or death, assessed up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Plitidepsin+Dexamethasone | Dexamethasone
Number analyzed (Participants) | 171 | 84
percentage of participants | 29.8 [23.1 to 37.3] | 1.2 [0.03 to 6.5]
Statistical Analysis 1: Comparison: Plitidepsin+Dexamethasone vs Dexamethasone; Test type: Superiority; p < 0.0001, Fisher Exact

17. Secondary Outcome: Overall Response Rate (Investigator Assessment) Excluding MR
Description: Very good partial response (VGPR) serum and urine M-protein detectable but not electrophoresis or >90% reduction in serum M-protein and urine M-protein <100 mg/24h Partial response (PR) ≥50% reduction in serum M-protein and 90% reduction in 24h urine M-protein or to <200 mg/24h. 50% reduction in size of any soft tissue plasmacytomas
Time Frame: From the date of first documentation of response to the date of disease progression or death, assessed up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Plitidepsin+Dexamethasone | Dexamethasone
Number analyzed (Participants) | 171 | 84
percentage of participants | 11.7 [7.3 to 17.5] | 1.2 [0.03 to 6.5]
Statistical Analysis 1: Comparison: Plitidepsin+Dexamethasone vs Dexamethasone; Test type: Superiority; p = 0.0029, Fisher Exact

ADVERSE EVENTS:
Time Frame: From first infusion to 30 days after the last administration of trial drug and until their resolution, an average of 5 years
Description: Four patients were not treated after randomization in Plitidepsin+Dexamethasone due to 2 deaths, 1 patient refusal and 1 reason not specified. One patient was not treated after randomization in Dexamethasone due to patient refusal
Arm/Group | Plitidepsin+Dexamethasone | Dexamethasone
All-Cause Mortality (participants affected / at risk) | 126/167 | 74/83
Serious Adverse Events (participants affected / at risk) | 99/167 | 26/83
Other Adverse Events (participants affected / at risk) | 161/167 | 80/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plitidepsin+Dexamethasone (N=167) | Dexamethasone (N=83)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasmablastic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Asthenia (General disorders) | 4 (4) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1)
General physical health deterioration (General disorders) | 2 (2) | 1 (1)
Malaise (General disorders) | 2 (2) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 8 (8) | 1 (1)
Thrombosis in device (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Drug administration error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 7 (10) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 6 (12) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0)
Blood creatine phosphokinase MB increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 6 (9) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 3 (3) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (4) | 0 (0)
Hepatic enzyme abnormal (Investigations) | 1 (1) | 0 (0)
Troponin I increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Plasma cells increased (Investigations) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (4) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (5) | 3 (4)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0)
Paresis (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Quadriparesis (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (8) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 4 (4) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 2 (3) | 3 (3)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myopathy toxic (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 6 (7) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 2 (2)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (2) | 0 (0)
Escherichia sepsis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (2) | 1 (1)
Lung infection (Infections and infestations) | 2 (2) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 15 (18) | 3 (3)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 2 (2) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Sepsis (Infections and infestations) | 9 (9) | 2 (2)
Septic shock (Infections and infestations) | 4 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 2 (2)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium colitis (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plitidepsin+Dexamethasone (N=167) | Dexamethasone (N=83)
Hypertension (Vascular disorders) | 14 (17) | 5 (6)
Hypotension (Vascular disorders) | 16 (17) | 1 (1)
Alanine aminotransferase increased (Investigations) | 22 (48) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 11 (20) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 28 (41) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 15 (34) | 1 (1)
Weight decreased (Investigations) | 12 (13) | 1 (1)
Platelet count decreased (Investigations) | 7 (67) | 5 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 31 (42) | 9 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 (36) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 6 (8)
Anaemia (Blood and lymphatic system disorders) | 69 (203) | 34 (97)
Neutropenia (Blood and lymphatic system disorders) | 12 (26) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 15 (47) | 8 (15)
Headache (Nervous system disorders) | 18 (18) | 5 (6)
Asthenia (General disorders) | 32 (60) | 9 (11)
Chest pain (General disorders) | 9 (12) | 2 (2)
Fatigue (General disorders) | 55 (95) | 18 (22)
Oedema peripheral (General disorders) | 31 (45) | 5 (6)
Pyrexia (General disorders) | 32 (50) | 11 (14)
Insomnia (Psychiatric disorders) | 18 (23) | 10 (11)
Abdominal pain upper (Gastrointestinal disorders) | 16 (16) | 1 (1)
Constipation (Gastrointestinal disorders) | 21 (23) | 5 (7)
Diarrhoea (Gastrointestinal disorders) | 57 (80) | 8 (10)
Dyspepsia (Gastrointestinal disorders) | 9 (12) | 4 (5)
Nausea (Gastrointestinal disorders) | 76 (122) | 17 (19)
Vomiting (Gastrointestinal disorders) | 41 (57) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (18) | 15 (22)
Bone pain (Musculoskeletal and connective tissue disorders) | 12 (13) | 15 (17)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 21 (27) | 3 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 (14) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 30 (47) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 34 (40) | 5 (5)
Hypercalcaemia (Metabolism and nutrition disorders) | 8 (9) | 7 (11)
Hyperglycaemia (Metabolism and nutrition disorders) | 11 (16) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 19 (23) | 5 (5)
Nasopharyngitis (Infections and infestations) | 5 (5) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 14 (19) | 5 (5)
Urinary tract infection (Infections and infestations) | 12 (13) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review.

DOCUMENTS (2):
  • Study Protocol (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT01102426/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT01102426/SAP_001.pdf